CLINICAL TRIAL: NCT06129669
Title: Determining Critical Thresholds of Tissue Perfusion With ICG in Reconstructive Surgery
Brief Title: ICG Indocyanine Green in Reconstructive Surgery
Acronym: ICG-R
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Caroline Driessen, Plastic Surgeon, Amsterdam UMC, location VUmc
Other Study IDs: NL74852.029.21
Record Dates: First submitted 2023-10-11; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Surgery; Fluorescence
Keywords: Reconstructive surgery; Free flap; Pedicled flap; Debridement; Fluorescence imaging; Indocyanine green
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Debridement after radiotherapy: Debridement after radiotherapy
  Interventions: Drug: Indocyanine green
- Debridement after trauma: Debridement after trauma
  Interventions: Drug: Indocyanine green
- Reconstructive surgery using a fasciocutaneous flap: Reconstructive surgery using a fasciocutaneous flap
  Interventions: Drug: Indocyanine green
- Reconstructive surgery using a muscle flap: Reconstructive surgery using a muscle flap
  Interventions: Drug: Indocyanine green
- Reconstructive surgery using a osseous flap: Reconstructive surgery using a osseous flap
  Interventions: Drug: Indocyanine green
- Vaginaplasties: Vaginaplasties using a peritoneum flap or colon interposition
  Interventions: Drug: Indocyanine green
- Phalloplasties: Phalloplasties
  Interventions: Drug: Indocyanine green
- Finger replantation: Finger replantation
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Administration of ICG during surgery and recording of the fluorescence video to perform data analyses

SUMMARY:
The success or failure of a reconstruction is largely related to the vascularization of the operated area. Near infrared fluorescence (also near infrared fluorescence angiography, NIR FA) with ICG administration is an innovative technique to quantify tissue perfusion. Based on the results obtained in other subspecialties, NIR fluorescence appears to be a promising way to quantify tissue perfusion in reconstructive surgery. Fluorescence research has previously been used in the context of microsurgery and breast reconstructions using implants, but structural objective determinations are lacking. Our study is successful if we are able to determine a cut off value for the absolute or relative perfusion parameters.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Undergoing debridement and/or reconstructive surgery included in the aforementioned groups

Exclusion Criteria:

* allergy or hypersensitivity to sodium iodide, iodine, ICG or shellfish
* patients with hyperthyroidism and patients with autonomic thyroid adenoma
* pregnancy or lactation
* epilepsy
* severe liver failure
* renal failure with a GFR <60.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We include patients that undergo a surgical debridement and/or reconstruction. Each group consists of twenty patients.
  The debridement groups mainly consist of post-oncologic patients who have undergone radiotherapy (1A) and trauma patients (1B).
  Reconstructive groups include 2A Fasciocutaneous flaps 2B Osseous flaps 2C Muscle flaps 2D Vaginaplasties 2E Phalloplasties 2F Finger replantations
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Maximum perfusion intensity (Normal) | Once during the surgery
  1. Maximum perfusion intensity (Imax, units) in a normal vascularized reference frame
Maximum perfusion intensity (ROI) | Once during the surgery
  2. Maximum perfusion intensity (Imax, units) in a normal vascularized reference frame
Relative Perfusion | Once during the surgery
  Maximum perfusion intensity (Imax, units) in a normal vascularized reference frame / Maximum perfusion intensity (Imax, units) in a normal vascularized reference frame

SECONDARY OUTCOMES:
Tmax | Once during the surgery
  Time to reach maximum perfusion in region of interest (Tmax, sec)
Ingress | Once during the surgery
  Rate of increase in intensity from baseline to peak intensity (Ingress, units)
Egress | Once during the surgery
  Degree of decrease in intensity from peak to last measurement (Egress, units)
Lap Failure | Follow up at six weeks postoperative
  Quantified as I <5%; II 5-15%, III 15-50%, IV> 50%, V complete
Wound infection | Follow up at six weeks postoperative
  Defined as none, local wound treatment, antibiotics, or hospitalization.
Skin necrosis | Follow up at six weeks postoperative
  Defined as none, partial thickness, and full thickness.
Delayed union | Follow up at six and twelve months postoperative
  Radiologic examination (Xray or CT) concluding on the presence of delayed union after 6 months or non-union after 12 months
Relative Perfusion before and after tissue transfer | Twice during the surgery
  Maximum perfusion intensity (Imax, units) in the same reference frame after tissue transfer / Maximum perfusion intensity (Imax, units) in a reference frame before tissue transfer

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Driessen, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

REFERENCES:
- [Derived] Van 't Hof LWP, Koster ITS, Van den Elzen RM, Bouman MB, Botman M, Driessen C. Quantitative Perfusion Assessment Using Indocyanine Green in Lower Extremity Perforator Flaps. Surg Innov. 2025 Oct;32(5):435-441. doi: 10.1177/15533506251339929. Epub 2025 May 19. PMID 40387116